CLINICAL TRIAL: NCT06559033
Title: Determine the Frequency of Variants in the GBA/PSAP Genes in Patients With Multiple Myeloma (MM) or Monoclonal Gammopathy of Undetermined Significance (MGUS)
Brief Title: Determine the Frequency of Variants in the GBA/PSAP Genes in Patients With MM or MGUS
Acronym: GAMY
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/0430/OB; 2022-A00306-37 (Registry Identifier: French Minister)
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-08

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Myeloma Multiple
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA (DeoxyriboNucleic Acid) extraction for sequencing of beta-GlucocereBrosidAse (GBA) and ProSAPosin (PSAP) genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Multiple myeloma (MM) patient group: patients with multiple myeloma (MM) (defined by a clonal proliferation of tumour plasma cells (>10%), the presence of a monoclonal peak in the serum or urine (excluding non-secretory myeloma) and organ damage secondary to bone marrow invasion)
  Interventions: Biological: Evaluation of the presence and number of mutated alleles of the GBA/PSAP genes in patients with MM or MGUS
- Monoclonal gammopathy of undetermined significance (MGUS) patient group: patients with MGUS (defined as bone marrow plasmacytosis of less than 10%, associated with a monoclonal protein of less than 30g/L and no clinical involvement)
  Interventions: Biological: Evaluation of the presence and number of mutated alleles of the GBA/PSAP genes in patients with MM or MGUS
- Control group: patient with no pathology under study relating to the project
  Interventions: Biological: Evaluation of the presence and number of mutated alleles of the GBA/PSAP genes in patients with MM or MGUS

INTERVENTIONS:
Biological: Evaluation of the presence and number of mutated alleles of the GBA/PSAP genes in patients with MM or MGUS — Estimation of the frequency of variants in the PSAP/GBA genes in patients with MM or MGUS, then comparison with a reference frequency from databases such as the Exome Aggregation Consortium, the Exome Sequencing Project, the 1000 Genomes Project and the dbSNP.
  Other Names: Evaluation of plasma concentrations of LGL1 in patients with MM or MGUS compared to controls; Evaluation of the % Reactivity of plasma immunoglobulins from patients with MM or MGUS towards LGL1

SUMMARY:
No effective specific treatment is currently available for the management of Multiple Myeloma (MM) and Monoclonal Gammopathy of Undetermined Significance (MGUS). A better understanding of the pathophysiological mechanisms would make it possible to propose treatments specifically targeting the deregulated pathways.

DETAILED DESCRIPTION:
This study will characterise the links between rare diseases and complex, chronic diseases. Metabolism can be visualised as a complex network in which the various biomolecules represent metabolic nodes and are linked together by connections. The number of connections at a node influences the effect of that biomolecule on the metabolic network(s) as a whole. If a biomolecule has a large number of connections, altering a metabolic pathway involving it will have an effect that will spread throughout the network. On the other hand, metabolic pathways with a high flux have a major impact on the homeostasis of the network. Thus, alteration of such a metabolic pathway cannot be without consequence: a major alteration could induce a rare hereditary metabolic disease with an early-onset clinic, whereas an alteration with a moderate effect could participate in the pathogenesis of complex diseases, and may open up new therapeutic prospects for these tumour pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with multiple myeloma (MM) (defined by clonal proliferation of tumour plasma cells (>10%), presence of a monoclonal peak in serum or urine (excluding non-secretory myeloma) and organ involvement secondary to bone marrow invasion) or with MGUS (defined as bone marrow plasmacytosis of less than 10%, associated with a monoclonal protein of less than 30g/L and no clinical involvement).
* Membership of a social security scheme
* Adult having read and understood the information letter and signed the consent form

Exclusion Criteria:

* Person deprived of liberty by an administrative or judicial decision or person placed under court protection / sub-guardianship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with multiple myeloma (MM), 100 patients with monoclonal gammopathy of undetermined significance (MGUS), 100 controls with plasma samples available
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-10-02 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of variants in the GBA/PSAP genes in patients with MM or MGUS | inclusion (one day)
  The main aim of the research is to determine the frequency of variants in the GBA/PSAP genes in patients with MM or MGUS.

SECONDARY OUTCOMES:
Plasma concentrations of LGL1 in patients with MM or MGUS | inclusion (one day)
  Compare the plasma concentration of LGL1 in MM and MGUS patients versus control individuals
Reactivity of monoclonal antibodies in MM and MGUS patients | inclusion (one day)
  Assess the % (proportion of patients with reactivity (% reactivity greater than 0) and those without (% reactivity equal to 0)) of reactivity of monoclonal antibodies from MM and MGUS patients to LGL1

IPD SHARING:
Plan to Share IPD: No